CLINICAL TRIAL: NCT07222293
Title: Assessment of 'DRISTi' as an Automated Diabetic Retinopathy Screening Tool in Diabetic Populations
Brief Title: Assessment of AI Program 'DRISTi' as a Screening Tool
Status: Recruiting | Type: Observational
Sponsor: Artelus AI (Industry)
Responsible Party: Sponsor
Other Study IDs: 25-02-199
Record Dates: First submitted 2025-10-25; First posted 2025-10-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Retinopathy (DR)
Keywords: Artificial Intelligence; Ophthalmic Device; AI; Diabetic Retinopathy; Diabetes; DR; Screening; Online/Offline; Fundus Camera
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Fundus Image Grading — The image is graded by a fully automated AI device

SUMMARY:
A study will be conducted to demonstrate that DRISTi will correctly diagnose Diabetic Retinopathy (e.g., mtmDR, PDR, DME) in eyes of patients with diabetes. Participants who have been diagnosed with diabetes mellitus and meet the other inclusion/exclusion criteria will be invited to participate and will consent to have ophthalmic images taken. These images will be analyzed by DRISTi AI software and evaluated by an ophthalmic reading center. The results will be compared, and a statistical analysis will be completed to ensure statistical significance in the outcomes thus proving DRISTi is an effective DR diagnosis tool.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to sign and date the informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age (≥)21 years of age or older
4. Diagnosed with diabetes mellitus as per criteria established by the World Health Organization (WHO) or the American Diabetes Association (ADA)

   1. Hemoglobin A1c (HbA1c) ≥ 6.5%
   2. Fasting Plasma Glucose (FPG) ≥ 126 mg/dL (7.0 mmol/L)
   3. Symptoms of hyperglycemia or hyperglycemic crisis with a random plasma glucose (RPG) ≥ 200 mg/dL (11.1 mmol/L)

Exclusion Criteria:

1. Persistent visual impairment in one or both eyes;
2. History of macular edema or retinal vascular (vein or artery) occlusion;
3. History of ocular injections, laser treatment of the retina, or intraocular surgery other than cataract surgery without complications;
4. Subject is contraindicated for fundus photography (for example, has light sensitivity);
5. Subject has contraindications for mydriatic medications or is unwilling or unable to dilate;
6. Subject is currently enrolled in an interventional study of an investigational device or drug for the same condition; or
7. Subject has a condition or is in a situation which in the opinion of the Investigator, might confound study results, may interfere significantly with the subject's participation in the study, or may result in ungradable clinical reference standard photographs
8. Subject falls into one of the below categories:

   * Adults unable to consent (individuals w/ impaired decision-making capacity)
   * Individuals who are not yet adults (infants, children, teenagers)
   * Pregnant women
   * Prisoners

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be referred from primary care clinics and ophthalmology clinics in North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-11-23 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI Grade | From time of arrival to completion of diagnostic tests, up to 8 hours
  AI generated image grades are directly compared to a Human generated image grade

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Jindal, MD, Principal Investigator — New Century Ophthalmology
Locations (2):
- United States (2):
  - New Century Ophthalmology - Oxford, Oxford, North Carolina
  - New Century Ophthalmology - Raleigh, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No
resource constraints